CLINICAL TRIAL: NCT03800979
Title: Effectiveness and Safety of Tofacitinib in Patients With Extensive and Recalcitrant Alopecia Areata
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Dermatology, Thailand (Other Government)
Responsible Party: Principal Investigator, Chinmanat Lekhavat, Assistant Director of Institute of Dermatology, Institute of Dermatology, Thailand
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB/IEB 004/2562
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Alopecia Areata
Keywords: Alopecia areata; Alopecia universalis; Alopecia totalis; Tofacitinib; JAK inhibitor
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis | interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: This is a Cohort study which all recruited volunteers will receive Tofacitinib for total of 24 weeks. The 19 volunteers are mixed male and female Thais who suffer from severe AA over 50% of the entire scalp.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tofacitinib (Experimental): All participants will take Tofacitinib 5 mg twice daily for 24 weeks to treat extensive and recalcitrant alopecia areata.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Tofacitinib is an oral medicine in Janus kinase inhibitor 3 group which has been approved by FDA in treating Rheumatoid Arthritis. It has ability to inhibit nerve signal Interferon-ɣ and Interleukin-15 between white blood cell(WBC) and the nucleus of hair follicle cell causing the production of WBC type CD8+NKG2D+ T cell to slow down which this type of WBC is one of the cause of hair loss.
  Other Names: Xeljanz

SUMMARY:
The objective of this study is to assess the safety and efficacy of Tofacitinib in treating patients with extensive and recalcitrant Alopecia Areata (AA), along with to evaluate the economic impact of the patients that may be from changing in their quality of life. There are patients with severe AA who may have little or no improvement from the treatment by diphenylcyclopropenone (DPCP) or topical steroid with minoxidil but instead having positive response from the treatment with Janus kinase(JAK) inhibitor such as Tofacitinib or Ruxolitinib. For the best of my knowledge, there was no previous study in using Tofacitinib to treat severe AA before in Thailand.

DETAILED DESCRIPTION:
Alopecia areata (AA) or spot baldness, is a condition in which hair falls off from areas of the body. It often happens on the scalp, causing a few bald spots and it may result in psychological stress even though people are generally healthy. AA is believed to be an autoimmune disease progressing from a breach in the immune privilege of the hair follicles that causes hair to fall out in small patches, it may remain unnoticeable until the patches eventually connect and then become noticeable. It can develop slowly, and also recur after years between occurrences.

By standard AA treatment guideline, DPCP is the first treatment protocol and may follow with anthralin or minoxidil. This oldy but goody treatment gives a good result of 75% in spotty hair loss and 25% in total baldness. The new invention of treatment has been introduced in the past 2 years by using JAK inhibitor, an oral medicine such as Tofacitinib and Ruxolitinib. This treatment gives a good outcome so far in this short period of time, 54-81.9% of patients had over 50% increase of hair grows over the original protocol. The theory is that JAK inhibitors would inhibit interferon-gamma and interleukin-15 signal between white blood cell and hair follicle which reducing the rate of destroying hair follicles.

The investigators propose the study to assess the safety and efficacy of Tofacitinib for extensive and recalcitrant AA and to evaluate the economic impact effecting the AA patients. Tofacitinib is an expensive medicine and needed to be taken up to 6 months to finish the course to have a best outcome so it is not a popular choice of AA treatment at present time unless it can show a promising result in recalcitrant AA.

ELIGIBILITY:
Inclusion Criteria:

* Thai volunteers age between 18 and 60 years old.
* Volunteers must be patients who suffer from severe AA more than 50% of the entire scalp.
* Volunteers must be patients who are able to complete the monthly treatment at least in the first 6 months.

Exclusion Criteria:

* Patients who suffer from other hair diseases such as: Telogen effluvium, Trichotillomania, Tinea capitis
* Patients who have other diseases that can have an impact on hair loss or temporary hair loss condition with in 6 months prior to the study such as: thyroid problems, liver disease, malnutrition, hearth disease, neurological disease, gastrointestinal disorders, sexually transmitted disease, cancer, psychiatric disease.
* Patients with AA who received treatment with either steroid, Anthralin or DPCP application within 1 month before the selection or patients who had oral or injection from steroid or other medication for hair loss treatment within 3 months before the selection.
* Woman with pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chinmanat Lekhavat, MD, Principal Investigator — Institute of Dermatology
Locations (1):
- Institute of Dermatology, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alkhalifah A, Alsantali A, Wang E, McElwee KJ, Shapiro J. Alopecia areata update: part II. Treatment. J Am Acad Dermatol. 2010 Feb;62(2):191-202, quiz 203-4. doi: 10.1016/j.jaad.2009.10.031. PMID 20115946
- [Background] Tosti A, Iorizzo M, Botta GL, Milani M. Efficacy and safety of a new clobetasol propionate 0.05% foam in alopecia areata: a randomized, double-blind placebo-controlled trial. J Eur Acad Dermatol Venereol. 2006 Nov;20(10):1243-7. doi: 10.1111/j.1468-3083.2006.01781.x. PMID 17062039
- [Background] Taylor CR, Hawk JL. PUVA treatment of alopecia areata partialis, totalis and universalis: audit of 10 years' experience at St John's Institute of Dermatology. Br J Dermatol. 1995 Dec;133(6):914-8. doi: 10.1111/j.1365-2133.1995.tb06925.x. PMID 8547044
- [Background] Liu LY, Craiglow BG, Dai F, King BA. Tofacitinib for the treatment of severe alopecia areata and variants: A study of 90 patients. J Am Acad Dermatol. 2017 Jan;76(1):22-28. doi: 10.1016/j.jaad.2016.09.007. Epub 2016 Nov 2. PMID 27816293
- [Background] Craiglow BG, Liu LY, King BA. Tofacitinib for the treatment of alopecia areata and variants in adolescents. J Am Acad Dermatol. 2017 Jan;76(1):29-32. doi: 10.1016/j.jaad.2016.09.006. Epub 2016 Nov 2. PMID 27816292
- [Background] Ibrahim O, Bayart CB, Hogan S, Piliang M, Bergfeld WF. Treatment of Alopecia Areata With Tofacitinib. JAMA Dermatol. 2017 Jun 1;153(6):600-602. doi: 10.1001/jamadermatol.2017.0001. PMID 28355451
- [Background] Divito SJ, Kupper TS. Inhibiting Janus kinases to treat alopecia areata. Nat Med. 2014 Sep;20(9):989-90. doi: 10.1038/nm.3685. PMID 25198048
- [Result] Alkhalifah A, Alsantali A, Wang E, McElwee KJ, Shapiro J. Alopecia areata update: part I. Clinical picture, histopathology, and pathogenesis. J Am Acad Dermatol. 2010 Feb;62(2):177-88, quiz 189-90. doi: 10.1016/j.jaad.2009.10.032. PMID 20115945

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Nineteen participants who met the inclusion criteria were enrolled and received 10 mg/day oral tofacitinib.
Groups:
- Tofacitinib: All participants will take Tofacitinib 5 mg twice daily for 24 weeks to treat extensive and recalcitrant alopecia areata.
  Tofacitinib: Tofacitinib is an oral medicine in the Janus kinase inhibitor 3 groups which FDA has approved in treating Rheumatoid Arthritis. It can inhibit nerve signal Interferon-ɣ and Interleukin-15 between white blood cell(WBC) and the nucleus of hair follicle cell causing the production of WBC type CD8+NKG2D+ T cell to slow down which this type of WBC is one of the causes of hair loss.
Period: Overall Study
Arm/Group | Tofacitinib
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Tofacitinib: All participants will take Tofacitinib 5 mg twice daily for 24 weeks to treat extensive and recalcitrant alopecia areata.
  Tofacitinib is the Janus kinase inhibitor, which FDA has approved for Rheumatoid Arthritis. It can inhibit nerve signal Interferon-ɣ and Interleukin-15 between white blood cell(WBC) and the nucleus of hair follicle cell causing the production of WBC type CD8+NKG2D+ T cell to slow down which this type of WBC is one of the causes of hair loss.
Arm/Group | Tofacitinib
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.68 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 19
Region of Enrollment [Count of Participants; unit: Participants]
  Thailand | 19
Baseline SALT score [Mean (Standard Deviation); unit: score] — Baseline SALT (Severity of Alopecia Tool) score is the percentage of hair loss. The total SALT score is measured 0-100%, with higher values representing greater hair loss.
  score | 95.11 (14.24)

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders vs Non-Responders Using SALT Score
Description: The Severity of Alopecia Tool (SALT) is a measurement procedure used by dermatologists to determine the percentage of scalp hair loss. The SALT system divides the scalp into 4 areas: Top has 4 sections of 10% total are 40%, back has 4 sections of 6% total are 24% and the 2 sides, left and right, each has 2 sections of 4% and 2 sections of 5% total of 18% and 36% combined. In the beginning, the area of hair loss would be measured by checking each area for hair loss and determining the bald spots combined per SALT scale then keeping the record as SALT baseline (SALT). The total SALT score is measured 0-100%, with higher values representing greater hair loss.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 19
Participants
  Responders (SALT score improved >=50%) | 9
  Non-responders (SALT score improved < 50%) | 10

2. Secondary Outcome: Side Effects From Tofacitinib
Description: Patients came back for follow-up every month during a total of 24 weeks of treatments and at weeks 28,36 and 48.
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 19
participants
  Dyslipidemia | 9
  Upper respiratory tract infection | 6
  Tuberculosis | 1
  Myalgia | 1
  Acne | 2
  Weight gain | 1
  Constipation | 1

ADVERSE EVENTS:
Time Frame: Patients came back for follow-up every month during a total of 24 weeks of treatments and at weeks 28,36 and 48.
Arm/Group | Tofacitinib
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 9/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tofacitinib (N=19)
Intestinal tuberculosis (Gastrointestinal disorders) | 1 (1) — Ileal tuberculosis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tofacitinib (N=19)
Dyslipidemia (Metabolism and nutrition disorders) | 9 (9) — Dyslipidemia (mild)
Upper respiratory tract infection (Infections and infestations) | 6 (6) — Upper respiratory tract infection such as common cold
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Myalgia
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Weight gain (Metabolism and nutrition disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT03800979/Prot_SAP_000.pdf